CLINICAL TRIAL: NCT02938403
Title: In Vivo Experience With NRT to Increase Adherence and Smoking Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Karen Cropsey, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA039678 (NIH); R01DA039678 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2025-04-07 (Actual); Status verified 2024-05

CONDITIONS: Smoking Reduction or Abstinence
MeSH Terms: conditions — Smoking Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In vivo group (Experimental): Those who receive in vivo counseling and Nicotine Replacement Therapy (NRT)
  Interventions: Behavioral: In vivo counseling
- Controls (Active Comparator): Standard smoking cessation counseling and Nicotine Replacement Therapy (NRT)
  Interventions: Behavioral: Standard Smoking Cessation Counseling

INTERVENTIONS:
Behavioral: In vivo counseling — Participants in the intervention group will receive 4 in session nicotine replacement therapy and counseling focused on their experience of using NRT, including positive experiences, side effects and smoking cessation expectancies. They will also received nicotine replacement therapy (nicotine lozenge and patch) to use for smoking cessation.
  Arms: In vivo group
Behavioral: Standard Smoking Cessation Counseling — Participants will receive 4 sessions of standard behavioral counseling to address their smoking. In addition, participants will received nicotine replacement therapy (Nicotine lozenge and patch) to use for smoking cessation.
  Arms: Controls

SUMMARY:
This is a study to determine the efficacy of a smoking cessation intervention (nicotine replacement therapy (NRT) and counseling) done in a systematized manner with participants recruited from the UAB Substance Abuse Program. The definition of In Vivo experience is: use of the NRT medication during the session using specialized counseling focused around their experience of using NRT, including how the use of NRT may help them quit smoking, side effects, and smoking cessation expectancies. In this study those in the In Vivo group will put the patch on during Session 1 and given nicotine gum in Session 2 and will discuss the experience of wearing the patch or chewing the gum while they are in session. The control group will not put on the patch or chew gum during the sessions but will be given standard counseling regarding quitting smoking.

DETAILED DESCRIPTION:
Aim 1: Compare the efficacy of an In Vivo experiential intervention to a standard treatment control group for smoking cessation. The goal of this aim will be to compare the rates of point prevalence abstinence at the 6 month post-intervention follow-up. It is expected that smokers who receive the behavioral experience of the NRT In Vivo intervention will have higher rates of abstinence at the 6 month follow-up compared to the control group. Aim 2: Compare medication adherence between groups over the 12 week intervention. The goal of this aim is to determine the impact of the In Vivo behavioral experience intervention on promoting medication adherence to NRT. It is expected that individuals in the In Vivo NRT group will have better medication adherence relative to control participants. Exploratory: Examine moderators and mediators of the experimental intervention on smoking abstinence. The goal of this aim is to explore whether demographic and smoking characteristics (e.g., sex, race, nicotine dependence, motivational status, legal charges) moderate the effect of treatment on abstinence after 12 weeks of treatment and 6-month follow-up. In addition, we will look at changes in expectancies about NRT, medication adherence, and withdrawal symptoms to determine if these changes mediate the relationship between the experimental intervention and smoking abstinence.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age,
* Under criminal justice supervision and expecting to remain under supervision for 9 months,
* Smoked at least 5 cigarettes per day for the last 12 months,
* Expire carbon dioxide (CO)> 10 ppm.
* Must be able to read and speak English.
* Women of child-bearing potential must be using adequate birth control.

Exclusion Criteria:

* Pregnant or breastfeeding women,
* Non-English speaking,
* Living in an restricted environment that does not allow smoking,
* Known sensitivity to nicotine replacement or allergy to adhesive used in nicotine patches,
* Cognitive impairment or major untreated mental illness that interferes with the informed consent process,
* Within 6 months post-myocardial infarction or untreated severe angina,
* Latex allergy,
* Daily or exclusive use of other tobacco products (e.g. cigars, e-cigarettes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | 6 months
  Smoking abstinence will be defined at 6 months as a CO< or equal to 3ppm and no smoking over the last 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Substance Abuse, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hawes ES, Mildrum Chana S, Faust A, Baker JC, Hendricks PS, Azuero A, Lahti AC, Carpenter MJ, Cropsey KL. In vivo Experience With NRT to Increase Adherence and Smoking Abstinence Among Individuals in the Criminal Legal System: Study Protocol for a Randomized Clinical Trial. Front Psychiatry. 2022 Jun 21;13:886680. doi: 10.3389/fpsyt.2022.886680. eCollection 2022. PMID 35800020